CLINICAL TRIAL: NCT06314984
Title: Effectiveness of Jet Injector Local Anesthesia Versus Conventional Technique in Primary Molars Pulpotomy
Brief Title: Jet Injectors Versus Conventional Anesthetic Technique in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Elbadry, Asistant lecturer at pediatric dentistry department, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A10040521
Record Dates: First submitted 2024-02-19; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Anesthesia
Keywords: Jet injector; Needle; Comfort-in; Pain perception; Needleless; Pediatric Dentistry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I A (Conventional neddle syringe) (Active Comparator): The injection was done in the mandible by the conventional needle syringe [Inferior Alveolar Nerve Block].
  Interventions: Other: Group I A (Conventional needle syringe)
- Group I B (Conventional needle syringe) (Active Comparator): The injection was done in the maxilla by the conventional needle syringe [Infiltration].
  Interventions: Other: Group I B (Conventional needle syringe)
- Group II A (Comfort-in Jet Injector) (Experimental): The injection was done in the mandible by the needleless Comfort-in jet injector [Inferior Alveolar Nerve Block].
  Interventions: Device: Group II A (Comfort-in Jet Injector)
- Group II B (Comfort-in Jet Injector) (Experimental): The injection was done in the maxilla by the needleless Comfort-in jet injector [Infiltration].
  Interventions: Device: Group II B (Comfort-in Jet Injector)

INTERVENTIONS:
Other: Group I A (Conventional needle syringe) — The injection site was isolated using cotton roll and the topical anesthesia (Benzocaine 4%) was applied to the injection site and left for 3-5 minutes then the injection was done in the mandible by the conventional needle syringe [Inferior Alveolar Nerve Block].
  Arms: Group I A (Conventional neddle syringe)
Other: Group I B (Conventional needle syringe) — The injection site was isolated using cotton roll and the topical anesthesia (Benzocaine 4%) was applied to the injection site and left for 3-5 minutes then the injection was done in the maxilla by the conventional needle syringe [Infiltration].
  Arms: Group I B (Conventional needle syringe)
Device: Group II A (Comfort-in Jet Injector) — The injection site was isolated using a cotton roll and the topical anesthesia (Benzocaine 4%) was applied to the injection site and left for 3-5 minutes then the injection was done in the mandible by the needleless Comfort-in jet injector [Inferior Alveolar Nerve Block].
  Arms: Group II A (Comfort-in Jet Injector)
Device: Group II B (Comfort-in Jet Injector) — The injection site was isolated using cotton roll and the topical anesthesia (Benzocaine 4%) was applied to the injection site and left for 3-5 minutes then the injection was done in the maxilla by the needleless Comfort-in jet injector [Infiltration].
  Arms: Group II B (Comfort-in Jet Injector)

SUMMARY:
This clinical study was conducted to compare the needleless Comfort-in jet injector device and the conventional needle technique in terms of

1. Pain level during the administration of local anesthesia in children.
2. Their effectiveness during pulpotomy procedures in primary molars.

Whether comfort-in jet injector device will achieve sufficient anesthesia for the procedures undertaken during pulpotomy or not when compared to the conventional technique and the pain levels of both techniques during the anesthesia step.

DETAILED DESCRIPTION:
Cooperative healthy seventy-six children required pulpotomy treatment in primary molars aged 4 to 7 years with no previous dental local anesthetic experience, were recruited from the pediatric dental clinic, Faculty of Dentistry, Mansoura university. The patients' behavior was categorized as positive or definitely positive according to Frankl Behavior Scale. All children were divided randomly into two main groups (38 each), control group I (conventional needle) and experimental group II (Comfort-in). Then two sub-group were constructed, each consists of 19 children. Sub-group I A and II A (IANB) and sub-group I B and II B (maxillary infiltration), the chief complaint of the child was the main determinant for the side (right or left) to be injected. The jet injector technique was applied in 2 shots with (0.5 ml) each, to unify the dose with the conventional technique. After testing the anesthesia's profoundness, pulpotomy steps proceeded. Pain evaluation was set up according to two different subjective and objective scales, the WBFP and FLACC scales. All parents of the children included in this study answered a post-treatment questionnaire to measure the degree of satisfaction regarding the technique that was selected for his/her child. Data were collected, tabulated, and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Children who require local anesthetic injection for pulpotomy.
2. Cooperative children (positive or definitely positive on Frankel's scale).
3. Children who had no previous dental local anesthetic experience, to avoid the influence of a negative or positive memory.
4. Children who have been determined to be healthy and free of systemic diseases.
5. Children who do not have any contraindications for administering a local anesthetic agent.

Exclusion Criteria:

1. Children suffering from medical illness, neurosensory disturbances, and psychiatric disorders.
2. Children who could not comprehend the pain measures.
3. Children with emergencies and acute dental conditions.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Pain level during the administration of local anesthesia by Wong-Baker faces pain rating scale | During adminstration of local anesthesia procedures.
  The first scale is the Wong-Baker FACES Pain Rating scale, a subjective scale. The child was shown a collection of six cartoon faces with a variety of facial expressions, from a very happy face to a very sad face. The child was given a brief explanation of each face before being told to select the one that best reflected his or her feelings while receiving local anesthesia.
  Assessment of Scores:
  0= No Hurt 2= Hurts Little Bit 4= Hurts Little More 6= Hurts Even More 8= Hurts Whole Lot 10= Hurts Lots the description of the faces: Face 0 is very happy because he doesn't hurt at all. Face 1 hurts just a little bit. Face 2 hurts a little more. Face 3 hurts even more. Face 4 hurts a whole lot more. Face 5 hurts as much as you can imagine, although you do not have to be crying to feel this bad.
Pain levels during pulpotomy procedures steps by Wong-Baker faces pain rating scale | During the pulpotomy procedure.
  The first scale is the Wong-Baker FACES Pain Rating scale, a subjective scale. The child was shown a collection of six cartoon faces with a variety of facial expressions, from a very happy face to a very sad face. The child was given a brief explanation of each face before being told to select the one that best reflected his or her feelings during the steps of pulpotomy procedure.
  Assessment of Scores:
  0= No Hurt 2= Hurts Little Bit 4= Hurts Little More 6= Hurts Even More 8= Hurts Whole Lot 10= Hurts Lots the description of the faces: Face 0 is very happy because he doesn't hurt at all. Face 1 hurts just a little bit. Face 2 hurts a little more. Face 3 hurts even more. Face 4 hurts a whole lot more. Face 5 hurts as much as you can imagine, although you do not have to be crying to feel this bad.
Pain level during administration of local anesthesia in children by FLACC scale. | During adminstration of local anesthesia procedures.
  The second scale is theFace, Legs, Activity, Cry, and Consolability [FLACC scale], an objective scale, which was used to measure pain according to Face, Legs, Activity, Cry, and Consolability. An assistant was well-trained to measure and calibrate the FLACC scale during the administration of anesthesia. Each category receives a score between 0 and 2, giving a final score between 0 and 10.Assessment of Scores:
  0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Pain levels during pulpotomy procedures steps by FLACC scale. | During the pulpotomy procedure.
  The second scale is the Face, Legs, Activity, Cry, and Consolability [FLACC scale], an objective scale, which was used to measure pain according to Face, Legs, Activity, Cry, and Consolability. An assistant was well-trained to measure and calibrate the FLACC scale during the pulpotomy procedure. Each category receives a score between 0 and 2, giving a final score between 0 and 10.Assessment of Scores:
  0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University., Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No